CLINICAL TRIAL: NCT05944367
Title: The Use of Breath Volatile Organic Compounds (VOCs) in Early Detection of Acute Pulmonary Exacerbations in Cystic Fibrosis
Brief Title: The Use of Breath Volatile Organic Compounds in Early Detection of Acute Pulmonary Exacerbations in Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 20/PR/0175
Record Dates: First submitted 2023-06-14; First posted 2023-07-13 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a single-centre, prospective observational cohort study assessing the potential utility of the Owlstone Medical "Breath Biopsy" in early diagnosis of pulmonary infections in patients with cystic fibrosis (CF). In cystic fibrosis pulmonary infections occur frequently and are associated with decline in lung function and disease progression, therefore a cornerstone of CF management is early identification and treatment of infections. "Breath Biopsy" is a non-invasive novel technology that has been trialled extensively in diagnosis of a variety of medical conditions with promising results. The technology is based the identification of a unique profile of organic compounds in exhaled breath of patients with a certain medical condition. Making the diagnosis of pulmonary infections in patients with CF is clinically challenging and at present relies on imprecise diagnostic tests, and generally requires attendance of patients to hospital or clinic for assessment. Ultimately, this research aims to assess the feasibility of incorporating "Breath Biopsy" into this diagnostic pathway with the advantages of both improving diagnostic certainty and potentially allowing in-home diagnosis of infections related to CF. Furthermore, identification of organic compounds implicated in CF infections will improve the understanding of why these infections occur, which to date remains an area that is poorly understood. Five patients with CF-related pulmonary infections admitted to the inpatient CF unit at the Royal Papworth Hospital will be enrolled, and use "Breath Biopsy" devices provided by Owlstone medical to collect breath samples from these patients in order to determine whether a unique organic compound profile can be identified in CF exacerbations.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Cystic Fibrosis based on genetic testing and/or sweat chloride levels
2. F508Del homozygous or heterozygous (F508Del with another severe CFTR mutation)
3. Age over 18 years
4. Able to provide written informed consent
5. Current exacerbation requiring inpatient or outpatient treatment at Royal Papworth Hospital.
6. Chronic infection with Pseudomonas aeruginosa, as defined as >50% of sputum culture or cough swabs being positive in the preceding 12 months
7. Baseline FEV1 30%-with no predicted upper limit

Exclusion Criteria:

1. Patients unable to provide written informed consent
2. Patients whose clinical status precludes use of the ReCIVA (mask) Breath Sampler due to oxygen dependency or tachypnoea
3. Patients who require admission to intensive care
4. Lung transplant recipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Cystic Fibrosis who attend Royal Papworth Cystic Fibrosis Centre
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
The accuracy of the Owlstone Breath Biopsy System to Detect Change in Volatile Organic Compounds During and After an Acute Pulmonary Exacerbation in Adults with Cystic Fibrosis, Measured by Mass Spectrometry Analysis of the Collected Breath Sample. | Change from baseline in Volatile Organic Compounds profile at day 1, 7 and 14 of an acute pulmonary exacerbation.
  Participants will have a breath biopsy taken by breathing into a fitted mask at the start, during, end of an acute pulmonary exacerbation requiring intravenous antibiotics.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Papworth Hospital, Cambridge, Cambridgeshire, United Kingdom